CLINICAL TRIAL: NCT04921748
Title: Destination Sequence Effect Modifications After a 4-week Rehabilitation Program in Parkinson's Diseases Patients
Brief Title: Neurorehabilitation of Sequence Effect in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Neurorehab in PD
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease; Freezing of Gait
Keywords: Movement disorders; Gait analysis; Hypokinesia; Basal ganglia; Functional indipendence
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Hypokinesia | interventions — Neurological Rehabilitation; Rehabilitation; Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD+FOG group: Patients affected by Parkinson's Disease with freezing of gait (PD+FOG group)
  Interventions: Procedure: Neurorehabilitation
- PD-FOG group: Patients affected by Parkinson's Disease without freezing of gait (PD+FOG group)
  Interventions: Procedure: Neurorehabilitation

INTERVENTIONS:
Procedure: Neurorehabilitation — All patients will be treated with an in-hospital rehabilitation program focused on the rehabilitation of gait disorder in PD with 90-minute daily sessions, 6 days a week (Monday through Saturday) for four weeks. The rehabilitation treatment includes passive, active-assisted, and active exercises, isotonic and isometric exercises for the major muscles of the limbs and trunk, cardiovascular warm-up exercises, muscle stretching exercises for functional purposes, balance training exercises, specific motor exercise for hypokinesia, and 45 minutes of overground gait training delivered without devices or cueing The rehabilitation program is the same in PD patients with and without FOG.
  Other Names: Rehabilitation; Physical therapy

SUMMARY:
The sequence effect (SE), defined as a reduction in amplitude of repetitive movements, is a common clinical feature of Parkinson's disease (PD), being a major contributor to freezing of gait (FOG). During walking, SE manifests as a step-by-step reduction in step length when approaching a turn or gait destination (dSE). The investigators studied the effect of a 4-week rehabilitation program on the destination sequence effect in patients affected by Parkinson's disease with and without Freezing of Gait. All subjects were evaluated with inertial gait analysis for dSE recording.

DETAILED DESCRIPTION:
Gait impairment and freezing of gait (FOG) represent common and disabling symptoms of Parkinson's disease (PD). The antiparkinsonian therapy positively modulates a subset of gait parameters, such as speed of gait and stride length, while its impact on FOG is limited. Growing evidence supports the efficacy of neurorehabilitation in the treatment of PD across all phases of the disease. In the last years, the advent of reliable wearable devices has prompted the widespread study of several parameters of the parkinsonian gait in both clinical and research settings.

The sequence effect (SE), defined as a reduction in amplitude of repetitive movements, is a common clinical feature of several tasks of patients affected by PD, being identifiable in early as well as advanced stages of the disease. During walking, SE manifests as a step-by-step reduction in step length when approaching a turn or gait destination (destination sequence effect - dSE). SE is specifically pronounced in PD patients affected by FOG, and it arises immediately before a FOG episode induced by a turning or a dual-task.

SE may be acutely modulated by several rehabilitative strategies such as split-belt treadmill and reinforcement of visual cues, but not by repetitive transcranial magnetic stimulation (rTMS), antiparkinsonian drugs administration, and attention strategies did not influence the SE, the evidence on the role of neurorehabilitation on gait SE improvement and retention is extremely scarce.

The investigators plan to enroll 43 subjects according to sample size calculation. Patients will be divided into two groups: patients with freezing of gait (FOG) and without FOG. The subjects will be divided into two groups: 1) patients with freezing of gait (PD+FOG), or 2) patients without freezing of gait (PD-FOG). FOG phenotype is defined as: a score between 1 and 4 at either item "2.13 Freezing" or item "3.11 Freezing of gait" of the Unified Parkinson Disease Rating Scale (UPDRS).

All patients will be treated with a standardized 4-week rehabilitation in-hospital program. At hospital admission (T0), patients who fulfill inclusion/exclusion criteria will be tested with instrumental gait analysis and administration of a set of the following clinical scales: rating of PD related motor disability with the Unified Parkinson's Disease Rating Scale - part III (UPDRS-III); rating of functional independence as measured through the Functional Independence Measure (FIM); and rating of dependence in activity of daily living according to Barthel Index.

After that, patients will be treated with 90-minute daily rehabilitative sessions, 6 days a week (Monday through Saturday) for four weeks (passive, active-assisted, and active exercises, isotonic and isometric exercises for the major muscles of the limbs and trunk, cardiovascular warm-up exercises, muscle stretching exercises for functional purposes, balance training exercises, specific motor exercise for hypokinesia, and 45 minutes of overground gait training delivered without devices or cueing). The rehabilitation program will be the same in PD+FOG and PD-FOG groups. At the end of the rehabilitation program (T1), the patients will complete the study procedure with a second instrumental gait analysis evaluation and the administration of the same set of clinical scales. No modifications of the drug regimen were allowed during the study.

The gait analysis will be performed with wearable, wireless, inertial system, secured to the back of the patients between L5 and S1 vertebrae. All subjects will be recorded in the morning (between 9:00 a.m. and 11:00 a.m.) and in the ON condition. The investigators plan to record a walk, at a comfortable pace, of 20 meters. The subjects will stop independently at the end of the 20-meter pathway, clearly marked by a straight line on the ground. Gait assessments with episodes of freezing of gait or pauses will be discrded. For each subject, three optimal performed gait assessments will be recorded. Regarding gait parameters the investigators will record: speed (m/s), cadence (steps/minute), stride length (meter), step length (meter), stride duration (second), single support, double support, swing duration, stance duration (percentage stride distribution). The destination Sequence Effect (dSE) will be computed as a regression slope (β) of step length according to a previously described and validated methodology where step length is plotted against step number. Briefly, the length of the last six steps ahead of the final stride are plotted against the step number, and the linear regression slope (β) will represent a measure of dSE. In addition, the intercept (I) of the regression curve will be used as an indirect measure of gait hypokinesia. For each group, the relationship between gait hypokinesia and sequence effect is expressed by the function of the linear regression as follow: y = β (x) + I.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Hoehn and Yahr stage between I and IV
* Mini-Mental State Examination score above 24.

Exclusion Criteria:

* Major psychiatric or other neurological conditions,
* Rheumatological diseases
* Ophthalmic diseases
* Orthopedic diseases
* Ongoing or previous treatment with neuroleptic drugs
* Patients with deep brain stimulation
* Any change in dose or regimen of the anti-parkinsonian therapy in the last month before enrolment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by Idiopathic Parkinson's disease with and without freezing of gait to be consecutively enroll among those attending the Neurorehabilitation Department of the IRCCS Mondino Foundation (Pavia, Italy)
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Destination sequence effect (dSE) modifications | Change from baseline (T0) to four weeks (T1)
  Using an inertial gait analysis we will explore the modifications of destination sequence effect in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program

SECONDARY OUTCOMES:
Between-group comparison of dSE | Baseline (T0)
  Comparison of destination Sequence Effect in PD patients with FOG vs. PD patients without FOG
Gait hypokinesia modifications | Change from baseline (T0) to four weeks (T1)
  Using an inertial gait analysis we will explore the modifications of intercept "I" in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program
Speed modifications | Change from baseline (T0) to four weeks (T1)
  Using an inertial gait analysis we will explore the modifications of speed (m/s) in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program
Cadence modifications | Change from baseline (T0) to four weeks (T1)
  Using an inertial gait analysis we will explore the modifications of cadence (steps/min) in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program
Stride duration modifications | Change from baseline (T0) to four weeks (T1)
  Using an inertial gait analysis we will explore the modifications of stride duration (s) in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program
Stride lenght modifications | Change from baseline (T0) to four weeks (T1)
  Using an inertial gait analysis we will explore the modifications of stride length (m) in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program
Stance modifications | Change from baseline (T0) to four weeks (T1)
  Using an inertial gait analysis we will explore the modifications of stance phase (%) in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program
Swing modifications | Change from baseline (T0) to four weeks (T1)
  Using an inertial gait analysis we will explore the modifications of Swing phase (%) in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program
Double support modifications | Change from baseline (T0) to four weeks (T1)
  Using an inertial gait analysis we will explore the modifications of double support (%) in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program
Single support modifications | Change from baseline (T0) to four weeks (T1)
  Using an inertial gait analysis we will explore the modifications of single support (%) in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program
Motor disability improvement | Change from baseline (T0) to four weeks (T1)
  We will explore the changes in motor disability as measured by Unified Parkinson Disease Rating Scale - part III (UPDRS-III) in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program
Functional Independence improvement | Change from baseline (T0) to four weeks (T1)
  We will explore the changes in functional independence as measured by Functional Independence Measure (FIM) in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program
Dependence in activity of daily living improvement | Change from baseline (T0) to four weeks (T1)
  We will explore the changes in dependence in activity of daily living as measured by barthel Index in PD patients with and without freezing of gait treated with a 4-week in-hospital rehabilitation program

CONTACTS AND LOCATIONS:
Overall Officials: Roberto De Icco, MD, Principal Investigator — IRCCS Mondino Foundation, Pavia
Locations (1):
- IRCCS Mondino Foundation, Pavia, Italy

REFERENCES:
- [Background] Kang SY, Wasaka T, Shamim EA, Auh S, Ueki Y, Lopez GJ, Kida T, Jin SH, Dang N, Hallett M. Characteristics of the sequence effect in Parkinson's disease. Mov Disord. 2010 Oct 15;25(13):2148-55. doi: 10.1002/mds.23251. PMID 20669182
- [Background] Cao SS, Yuan XZ, Wang SH, Taximaimaiti R, Wang XP. Transverse Strips Instead of Wearable Laser Lights Alleviate the Sequence Effect Toward a Destination in Parkinson's Disease Patients With Freezing of Gait. Front Neurol. 2020 Aug 12;11:838. doi: 10.3389/fneur.2020.00838. eCollection 2020. PMID 32903360